CLINICAL TRIAL: NCT02069171
Title: The Cross-sectional and Questionnaire Study of Pelvic and Lower Extremity Lymphedema After Treatment of Gynecological Disease
Brief Title: Cross-sectional and Questionnaire Study for Leg Lymphedema
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Myong Cheol Lim, Faculty, Center for Uterine Cancer, National Cancer Center, Korea
Other Study IDs: NCC_GO_2012_01_2; NCCNCS-12-565 (Other Grant/Funding Number: (South Korea) National Cancer Center , IRB)
Record Dates: First submitted 2013-05-31; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Gynecologic Cancer
Keywords: Lower extremity edema; Lower leg lymphedema; Lower leg edema; Lymphedema; Pelvic lymph node dissection; Gynecologic Cancer Lymphedema Questionnaire
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- early ovarian cancer group
- locally advanced cervical cancer group
- primary endometrial cancer group

SUMMARY:
The purpose of this study is to identify the incidence,feature,clinical significance for leg lymphedema after gynecologic cancer treatment.

DETAILED DESCRIPTION:
Medical records will reviewed. And all patients who met the inclusion criteria will contacted by a telephone call by a clinical research coordinator. The telephone interview questionnaire for Lower Extremity Edema (LEE) and gynecologic cancer lymphedema questionnaire (GCLQ) will t take approximately 20-30 min to complete. The questionnaire for LEE included onset, severity, location, duration, and management. Patients will also questioned concerning deep vein thrombosis to exclude other causes of LEE. LEE is defined as subjective edema of lower extremity based on patients' complaint. LLL is defined based on a clinical diagnosis of lymphedema by a physician.

ELIGIBILITY:
* Inclusion criteria

  1. the patient who gynecologic cancer treatment at National Cancer Center , Korea(2001~2011)
  2. no active cancer treatment at the moment
  3. available telephone communication
* exclusion criteria 1. The patient unlikely to comply with the protocol

<More information by cancer type>

* early ovarian cancer group Inclusion criteria were early stage epithelial ovarian cancer*, no active treatment, available telephone communication with patients, and ability and willingness to provide verbal informed consent.

  *early ovarian cancer (FIGO stage I and II) at National Cancer Center, Korea who underwent cytoreductive and staging surgery between January 2001 and December 2010
* locally advanced cervical cancer group patients with locally advanced cervical cancer who treatment at National Cancer Center, Korea between October 2001 and July 2007. Of 222 patients with locally advanced cervical cancer, 74 patients were underwent pretreatment laparoscopic surgical staging and 148 patients received radiotherapy . Women with locally advanced cervical cancer, no active treatment at survey, available telephone communication, and ability and willingness to provide verbal informed consent were considered to include in the current study.
* primary endometrial cancer group patients with endometrial cancer who underwent surgery, no active treatment at survey, available telephone communication, and ability and willingness to provide verbal informed consent were considered to include in the current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patient who gynecologic cancer treatment at National Cancer Center (2001~2011)
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Gynecologic Cancer Lymphedema Questionnaire | The study outcome measure will be assessed by telephone interview , one time.
  There are no more follow up except one time telephone interview.

CONTACTS AND LOCATIONS:
Overall Officials: Myong Cheol Lim, MD,PhD, Principal Investigator — National Cancer Center, Korea